CLINICAL TRIAL: NCT01442610
Title: Effects of Rasagiline on Sleep Disturbances in PD: A Single Center, Randomized, Double-blind, Placebo run-in, Polysomnographic Clinical Phase IV Trial
Brief Title: Effects of Rasagiline on Sleep Disturbances in Parkinson's Disease
Acronym: RaSPar
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TUD-RaSPar-051
Record Dates: First submitted 2011-09-23; First posted 2011-09-28 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Sleep Disturbances; Parkinsons's Disease
Keywords: Rasagiline; Sleep disorder; Parkinson's disease; Sleep Disturbances in patients with parkinsons's disease
MeSH Terms: conditions — Parasomnias; Sleep Wake Disorders; Parkinson Disease | interventions — rasagiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rasagiline (Experimental): Effect of Rasagiline on sleep parameters in PD Patients
  Interventions: Drug: Rasagiline
- Placebo (Placebo Comparator): Effect of placebo on sleep parameters in PD Patients
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rasagiline — Rasagiline tablets 1mg once daily for 8 weeks
  Other Names: Azilect
  Arms: Rasagiline
Drug: Placebo — Placebo 1tablet once daily for 8 weeks
  Arms: Placebo

SUMMARY:
As the MAO-B inhibitor rasagiline is able to improve motor skills it might have positive effects on sleep disruption by reducing nocturnal akinesia. As it was reported to cause only minor sleep disruption in PD Patients, it might be able to improve sleep architecture. The investigators thus study the effects of Rasagiline on sleep disturbances measured by polysomnographic (PSG) evaluation of sleep efficacy and PDSS-2. Secondary measures are other sleep variables measured by PSG, sleep quality and daytime sleepiness assessed by standardized scales as well as cognitive function, depression and QoL index.

DETAILED DESCRIPTION:
Sleeping disorders are very common in patients with Parkinson's Disease (PD). Mainly initiation and maintenance of sleep is disturbed, therefore many patients suffer from daytime sleepiness and sleep attacks. Polysomnographic studies showed increased sleep fragmentation and frequent awakenings, increased amount of wakefulness during time in bed as well as reduced sleep efficacy and deep sleep time. In addition, increased sleep latency, REM-latency and decreased amounts of REM sleep were documented.

PD patients also suffer from primary sleep disorders like sleep disordered breathing and especially REM sleep behaviour disorder (RBD)and periodic limb movements in sleep (PLMS).

Not only neurochemical changes affecting cholinergic and monoaminergic systems, nocturnal hypokinesia and rigidity and painful dystonia due to the disease itself, but also medication side effects lead to impaired sleep-wake-control and reduced REM sleep.

Although levodopa medication and dopamine agonists reduce nocturnal hypokinesia and therefore improve insomnia they also have a potential impact on daytime sleepiness and are able to cause sleep disruption. The impact of dopaminergic therapy is complex showing biphasic effects with increased wakefulness and decreased REM-sleep frequency via stimulation of dopamine D1 receptors whereas low doses promote sleep via dopamine D2 receptors. In addition, acting of dopamine agonists via dopamine D3 receptors might be responsible for daytime sleepiness and sleep attacks.

However, as stimulation of the subthalamic nucleus improves mainly motor skills but also shows an important increase in sleep duration and quality, it could be suggested that by decreasing nocturnal hypokinesia improvement in sleep quality can be achieved.

Rasagiline mesylate was developed as a selective and irreversible MAO-B- inhibitor which is - unlike Selegiline - not metabolized to amphetamine derivates which are found to be partly responsible for negative effects on RBD and REM-sleep as well as sleep efficacy. Rasagiline is able to delay the need for initiating dopaminergic therapy, improves motor function in early and moderate to advanced PD and was shown to exhibit neuroprotective potential.

As different mechanisms of dopaminergic medication on different dopamine receptors are still not fully elucidated and in contrast to selegiline no side effects due to development of amphetamine derivates need to be taken into consideration, this study is to aim at evaluating the effects on sleep and daytime sleepiness of treatment with Rasagiline mesylate.

As Rasagiline is able to improve motor skills it might have positive effects on sleep disruption by reducing nocturnal akinesia. As it was reported to cause less sleep disruption in PD Patients than placebo it might be able to improve sleep architecture. Until now no clinical trial using polysomnographic techniques was performed to evaluate the effects of Rasagiline on sleep.

To study the effects of Rasagiline on sleep disturbances measured by polysomnographic (PSG) evaluation of sleep efficacy and PDSS-2.

Secondary measures are other sleep variables measured by PSG. In addition, sleep quality and daytime sleepiness assessed by standardized scales as well as cognitive function, depression indices and QoL index are measured.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients
* Age from 50 to 85 years
* Definite Parkinson's disease according to UK brain bank criteria
* Hoehn & Yahr I-III
* Relevant sleep disturbance (> 5 point in PSQI)
* Patient must be able to complete questionaires
* Stable antiparkinsonian medication for at least 4 weeks prior to screening
* Antiparkinsonian medication should be stable 30 days prior to screening until 10 days after end of study
* Written informed consent

Exclusion Criteria:

* Overreaction/allergies to study drug or one of its components
* Pregnancy and/or lactation period
* Women with childbearing potential not practicing an acceptable method of contraception (Pearl-Index <1)
* Non-permitted medication within two weeks prior to study inclusion and during study: Hypnotics, Amantadine, MAO inhibitors, SSRIs, SNRIs, tricyclic and tetracyclic antidepressants, all neuroleptics except clozapine and quetiapine
* Non-permitted medication during study: CYP P450 1A2 inhibitors (a.e. Ciprofloxacin, Cimetidine, Clarithromycin, Erythromycin, systemic Estrogen, Fluvoxamine, Isoniazid, Ketoconazole, Levofloxacin, Norfloxacin, Mexiletine, Paroxetine, Propafenone, Zileuton, Disulfiram, Ginseng, grapefruit juice, Ephedrine).
* Planned participation or participation in another clinical trial during the last 4 weeks prior to screening and during the whole trial period
* Epilepsy or epileptic seizure in the history
* Significant renal or hepatic impairment
* Legal incapacity or limited legal capacity
* Dementia or other psychiatric illness that prevent from giving informed consent.
* Any clinically significant medical illnesses which interfere with capability to participate in study
* History of sleep related breathing disorder or severe OSAS as characterized by PSG (> 30 AHI)
* Severe Depression (BDI > 17)
* Known history of cardiac arrhythmias, angina pectoris, narrow angle glaucoma, residual urine caused by benign prostatic hyperplasia, pheochromocytoma
* Patients requiring elective surgery requiring general anaesthesia during study period

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-10; Primary Completion 2015-03 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in sleep efficacy | baseline and 8 weeks
  Change from baseline in sleep efficacy (% in time in bed (TIB) / sleep partial time (SPT)) in polysomnography at 8 weeks
Change in PDSS-2 | Baseline and 8 weeks
  Change from baseline in sleep quality at 8 weeks

SECONDARY OUTCOMES:
Change in other sleep parameters | baseline and 8 weeks
  Change from baseline in sleep parameters e.g. portion of REM-sleep (%), portion of slow wave sleep (%), portion of light sleep (%), sleep latency (min), REM-sleep latency (min) in polysomnography at 8 weeks
Electrocardiography | baseline and 8 weeks
  Number of participants with adverse events
Laboratory parameter | baseline and 8 weeks
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Storch, MD, Principal Investigator — Dresden University of Technology, Dept. of Neurology
Locations (1):
- Dresden University of Technology, Dept. of Neurology, Dresden, Germany